CLINICAL TRIAL: NCT06891469
Title: Effects of an Acute High Dose of Caffeine on Physiological Responses and Performance During a Strength-Focused CrossFit® Workout: a Randomized, Double - Blinded, Crossover Study
Brief Title: Effects of an Acute Dose of Caffeine on the Performance of CrossFit Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, ZOI KONIDARI, DIETICIAN-NUTRITIONIST, Democritus University of Thrace
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: DPTH/EHDE/18605/118
Record Dates: First submitted 2025-03-04; First posted 2025-03-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy, Young Adults; Athletic Performance
Keywords: caffeine; rating of perceived exertion; lactate; performance; high intensity functional training; CrossFit®
MeSH Terms: interventions — Biotin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine (Active Comparator): Consumption of 7.1 ±0.7 mg/kg of body mass of anhydrous caffeine (Pure Caffeine tablets by Myprotein), 60 minutes before the start of the specific CrossFit training program (four rounds of five exercises, 50 seconds exercise/10 seconds rest)
  Interventions: Dietary Supplement: Caffeine administration according to body mass (moderate intake- 7 mg/kg)
- Placebo (Placebo Comparator): Consumption of biotin (BIOTIN tablets by Myprotein) as placebo, 60 minutes before the start of the specific CrossFit training program (four rounds of five exercises, 50 seconds exercise/10 seconds rest). The volunteers received the same number of capsules that they received in caffeine condition
  Interventions: Dietary Supplement: Placebo (Biotin Capsules)

INTERVENTIONS:
Dietary Supplement: Caffeine administration according to body mass (moderate intake- 7 mg/kg) — This randomized, double-blind, crossover study aimed to investigate the acute effects of caffeine consumption on physiological responses and performance during a strength-focused CrossFit workout. Participants will consume either anhydrous caffeine (7.1 ± 0.7 mg/kg of body mass) or placebo, 60 minutes before a CrossFit workout aiming to perform as many repetitions as possible.
  Arms: Caffeine
Dietary Supplement: Placebo (Biotin Capsules) — Consumption of biotin (BIOTIN tablets by Myprotein) at the same time as caffeine.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial was to investigate the effect of an acute dose of caffeine on CrossFit performance in young, healthy male CrossFit athletes. The main questions it aimed to answer were whether an acute dose of caffeine, compared to placebo:

* Can improve performance in a specific CrossFit workout
* Leads to a reduction in the Rating of Perceived Exertion
* Leads to an increase in blood lactate concentration at the end of the workout

Participants had to:

* Complete two sessions of a specific CrossFit training program (four rounds of five exercises, 50 seconds of exercise/10 seconds of rest), 60 minutes after consuming either anhydrous caffeine (7.1 ± 0.7 mg/kg of body mass) or an equivalent amount of placebo, aiming to perform as many repetitions as possible.
* Report subjective perception of fatigue using the Borg scale at the end of each round.

DETAILED DESCRIPTION:
Preliminary measurements The preliminary measurements included anthropometry, body composition estimation, dietary and habitual caffeine consumption assessment. To assess habitual caffeine consumption, the volunteers were asked to answer a questionnaire through an interview, which investigated the typical consumption of specific caffeine-containing foods and beverages over the past month. Additionally, medical history information was collected through personal interviews.

Main tests Aerobic fitness and maximum heart rate were assessed using the 20-meter shuttle run at an indoor gymnasium. For each main session, the volunteers arrived at the gym having followed specific preparation instructions. Specifically, they were instructed to avoid intense exercise for 24 hours before the test, be hydrated, eat a carbohydrate-rich meal 3-4 hours earlier, avoid alcohol for 24 hours before the test, and refrain from energy drinks, supplements, or caffeine on the test day.

The two main tests were conducted at the same time of day and under similar environmental conditions for each volunteer. After being weighed, the volunteers took either caffeine or biotin capsules, and, 40 minutes later, they began warming up so that the training session would start 60 minutes after taking the supplement. Before the warm-up, blood lactate concentration was measured using the Lactate Scout 4 automatic lactate analyzer.

The volunteers executed five exercises (50 seconds on, 10 seconds off) for four rounds, aiming to perform as many repetitions as possible with the correct technique. The five exercises were push-ups, power cleans, front squats, sit-ups, and deadlifts. The power clean, front squat, and deadlift were performed with an external load of approximately 40%, 50%, and 60% of body weight, respectively.

Performance was defined as the total number of repetitions per round (i.e. the sum of repetitions in all exercises per round), as well as the number of repetitions performed in each exercise per round.

At the end of each round, the rating of perceived exertion (RPE) was recorded using the 6-to-20 Borg scale, and, one minute after the end of the workout, blood lactate concentration was measured again.

HR was monitored using a HR monitor (Polar H10) throughout the workout and averaged over each round.

Additionally, after completing the training sessions, the volunteers provided information about possible side effects (tachycardia, palpitations, feelings of anxiety/discomfort, headache, dizziness).

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 18-40
* At least 2 years of experience with CrossFit programs
* Free of any medical condition that prevents the participant from performing the exercises of the training program at maximum capacity

Exclusion Criteria:

* Consumption of caffeine and guarana supplements, unless were discontinued for at least two weeks before participating in the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
Performance During CrossFit® Workout | After 5, 10, 15 and 20 minutes of exercise
  Performance was defined as the total number of repetitions completed by the volunteers in the CrossFit program, the repetitions of all exercises per round, and the repetitions of each specific exercise per round.
Rating of Perceived Exertion during the CrossFit program | during the last 10 s of the 5th, 10th, 15th and 20th minute of exercise
  Each partictipant had to record the subjective perception of fatigue, using the Borg scale (6 to 20, with higher score meaning feeling of higher exertion), at the end of each round of CrossFit program
Blood lactate concentration | 1st measurement before the warm up and 2nd measurement one minute after the end of workout (i.e. after 20 min of exercise)
  Blood lactate concentration was measured using the Lactate Scout 4 automatic lactate analyzer (EKF Diagnostics) in two time points: before the warm-up for CrossFit program and one minute after the end of the workout

SECONDARY OUTCOMES:
Heart Rate | Heart rate was measured every 1 second of exercise. For analysis, heart rate was averaged over the following time ranges: 1-5 , 6-10 , 11-15 and 16-20 minutes of exercise
  Throughout the workout, heart rate was monitored using a heart rate monitor (Polar H10)
Aerobic fitness assessment | baseline (during the 2nd visit)
  Maximum oxygen consumption was estimated using the 20-meter shuttle run test from the number of shuttles completed at exhaustion.
Maximum heart rate measurement | Heart rate was continuously recorded during the test (every 1 s), until exhaustion. The highest heart rate at the time of exhaustion was recorded.
  Maximum Heart rate was determined during the 20-meter shuttle run test. Heart rate was continuously recorded using a heart rate monitor (Polar H10).

CONTACTS AND LOCATIONS:
Overall Officials: ILIAS SMILIOS, Professor, Study Director — Democritus University of Thrace; VASSILIS MOUGIOS, Professor, Study Director — Aristotle University Of Thessaloniki; GREGORY C. BOGDANIS, Professor, Study Chair — Gregory C. Bogdanis National and Kapodistrian University of Athens, School of Physical Education and Sport Science
Locations (1):
- Stefanos Karalis Indoors Facilities, Athens, Byron, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: The study diresctors, the study chair and those who will evaluate the article for publication
URL: https://doi.org/10.6084/m9.figshare.28426292

REFERENCES:
- [Background] Pickering C, Grgic J. Caffeine and Exercise: What Next? Sports Med. 2019 Jul;49(7):1007-1030. doi: 10.1007/s40279-019-01101-0. PMID 30977054
- [Background] Guest NS, VanDusseldorp TA, Nelson MT, Grgic J, Schoenfeld BJ, Jenkins NDM, Arent SM, Antonio J, Stout JR, Trexler ET, Smith-Ryan AE, Goldstein ER, Kalman DS, Campbell BI. International society of sports nutrition position stand: caffeine and exercise performance. J Int Soc Sports Nutr. 2021 Jan 2;18(1):1. doi: 10.1186/s12970-020-00383-4. PMID 33388079
- [Background] Claudino JG, Gabbett TJ, Bourgeois F, Souza HS, Miranda RC, Mezencio B, Soncin R, Cardoso Filho CA, Bottaro M, Hernandez AJ, Amadio AC, Serrao JC. CrossFit Overview: Systematic Review and Meta-analysis. Sports Med Open. 2018 Feb 26;4(1):11. doi: 10.1186/s40798-018-0124-5. PMID 29484512
- See also: Full data set of measurement performed in the study — https://doi.org/10.6084/m9.figshare.28426292
- Available data/document: Individual Participant Data Set: https://doi.org/10.6084/m9.fig — https://figshare.com — figshare